CLINICAL TRIAL: NCT06387017
Title: Prospective Multicenter Cohort Study to Validate Four Groups of Biomarkers for Assessing Lung Cancer Risk Among Patients With Atheromatous Cardiovascular Disease in a Screening Pathway
Acronym: BIOCEPTION
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RCAPHM22_0411
Record Dates: First submitted 2024-04-04; First posted 2024-04-26 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Smoking-related Pathology; Atheroma; Non-progressive Cancer > 5 Years; Lung Cancer
MeSH Terms: conditions — Plaque, Atherosclerotic; Lung Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- all patients (Other)
  Interventions: Diagnostic Test: blood sampling; Diagnostic Test: stool collection; Radiation: low dose CT scan

INTERVENTIONS:
Diagnostic Test: blood sampling — blood collection
Diagnostic Test: stool collection — stool collection
Radiation: low dose CT scan — low dose CT scan evaluation

SUMMARY:
Interventional study with minimal risks and constraints, with evaluation of the incidence of lung cancers by low-dose thoracic CT scan without injection of contrast medium, of the immunological, inflammatory and metabolic blood profile and of the microbiota; systematic proposal of smoking cessation for active smokers or assistance in maintaining cessation.

DETAILED DESCRIPTION:
This study aims to validate candidate biomarkers associated with the risk of lung cancer diagnosis among patients with atheromatous disease associated with smoking.

hese candidate biomarkers were identified from blood and stool samples taken from the PREVALUNG cohort (NCT03976804), comprising 512 patients with at least one smoking-related atheromatous disease who underwent a thoracic CT lung cancer screening pathway (1 single screening round, i.e. one CT scan and one year of follow-up) at the Marie Lannelongue Hospital - Groupe Hospitalier Paris Saint-Joseph (Le Plessis-Robinson). This screening pathway led to the diagnosis of 14 patients (3%) with lung cancer, over 70% of whom were early-stage (I or II) and could be managed curatively by minimally invasive surgery (unpublished results, presented at the World Congress Lung cancer in Singapore on September 10 and 11, 2023). A case-control study nested in the PREVALUNG cohort compared the biological profiles of patients with suspected lung cancers or nodules with those of patients without lung nodules. Around 15,000 biomarkers per case and control were analyzed by standard statistical methods (descriptive and logistic regression), partial least square method and machine learning after reduction of the number of variables.

By analyzing several types of variables linked to inflammation, immunity, blood metabolomics and stool metagenomics, these analyses identified 14 biomarkers divided into 4 groups of candidate biomarkers associated with the diagnosis of lung cancers the second cohort, PREVALUNG ETOILE (NCT05649046), was recruited at Marseille's Hôpital Nord, using the same intervention methods as PREVALUNG, but extending the inclusion criteria to other tobacco-related diseases (atheroma, but also chronic bronchitis and tobacco-related cancers in remission for more than 5 years), to people who would have been eligible in the prospective-randomized studies that have shown that lung cancer screening reduces lung cancer mortality (NLST and NELSON), and to people meeting the criteria of the North American recommendations. The aim of the PREVALUNG ETOILE study is to set up and evaluate a lung cancer screening care pathway at the APHM, using a biological blood and faeces collection identical to that of PREVALUNG. PREVALUNG ETOILE plans to include 160 participants in 2023 (160 have already been included as of September 20, 2023). A 5-month follow-up after the first screening round is planned for each participant. The total number of participants to be included in Europe is 2750. The number of participants to be included in the French BIOCEPTION cohort will therefore be a maximum of 2,750. APHM is coordinating data collection from the various European centers involved in the PREVALUNG BIOCEPTION study. Pr Tatiana Kouznetsova of KU Leuven (Belgium) is in charge of the statistical analysis of the data, in collaboration with APHM.

The PREVALUNG BIOCEPTION cohort was set up to validate biomarkers of risk of incident lung cancer at 2 years, as part of screening. These biomarkers will subsequently serve as therapeutic targets for the primary prevention of lung cancer. As part of the PREVALUNG EU project, a prospective randomized 8-arm study is planned to demonstrate the biological effect of drug interventions on the 4 classes of biomarkers that will have been validated (see PREVALUNG EU appendix).

This protocol is therefore part of a scientifically validated project funded by the European Commission for the validation of biological biomarkers and the primary prevention of lung cancer risk in patients with smoking-related atheromatous disease. External validation of biomarkers from a cohort of participants at risk of lung cancer without atheromatous disease or moderate or severe calcium score (some participants of PREVALUNG ETOILE or newly recruited) will initiate the extension of the validation and application of these biomarkers to non-atheromatous populations.

ELIGIBILITY:
Inclusion Criteria:

* 1- All PREVALUNG or PREVALUNG ETOILE participants
* 2- Active or former smokers who have smoked daily for at least 10 years and have either atheromatous disease (coronary, lower limb, supra-aortic trunk, aortic, visceral or upper limb arteries) or a moderate or high coronary calcium score*, **.

Inclusion criteria:

* Age 45- 75 years and
* Medical follow-up for smoking-related atheromatous pathology and
* daily smoking for at least 10 years prior to disease (for smoking, there are no quantitative criteria or withdrawal times)

  * visual coronary calcium score quantified by a radiologist on a chest CT scan.

    3- Individuals at risk of lung cancer without atheromatous disease or moderate or high calcium score being managed for a tobacco-related disease (chronic bronchitis or non-progressive cancer > 5 years) or with eligibility criteria for lung cancer screening (inclusion criteria in the NLST or NELSON studies or American recommendations)**.

Inclusion criteria :

* Age 45- 75 and
* Medical follow-up for a smoking-related pathology:
* chronic obstructive pulmonary disease / emphysema, or
* history of non-progressive cancer > 5 years, including ENT, lung, breast, cervix, excreto-urinary tract, bladder, esophagus, stomach, pancreas, liver, kidney, chronic myeloid leukemia.

and

- daily smoking for at least 10 years prior to the disease (for smoking, there are no quantitative criteria or withdrawal periods).

Or

Inclusion criteria in NLST :

* Age 55 - 74
* Cumulative smoking ≥ 30 pack-years
* active or weaned for less than 15 years Or

NELSON inclusion criteria :

* Age 50-75
* Smoking :
* > 15 cigarettes /D for more than 25 years or
* > 10 cigarettes /D for more than 30 years
* active smoking or cessation < 10 years Or

American recommendations :

* Age 50 - 80
* Smoking ≥20 PA

Exclusion Criteria:

* cancer history < 5 years (except carcinoma in situ of the uterine cervix, basal cell carcinoma of the skin, non-invasive urothelial carcinoma treated for curative purposes without CT lung surveillance, prostate cancer with unmeasurable PSA)
* symptoms of lung cancer (involuntary weight loss > 7 kg in 1 year, hemoptysis)
* known history of pulmonary nodule requiring specialized follow-up
* history of pulmonary fibrosis or pulmonary hypertension
* active pulmonary parenchymal infection
* severe cardiac or respiratory insufficiency (rest dyspnea)
* performance status (WHO) 2, 3 or 4
* patient not affiliated to the social security system (beneficiary or beneficiary's beneficiary)
* patient deprived of liberty
* patients under guardianship or trusteeship
* pregnant or breast-feeding women

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 750 (Estimated)
Dates: Start 2024-04-02 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
biomarker group validation | 51 months
  Sensitivity and specificity of each biomarker

SECONDARY OUTCOMES:
Describe changes in biomarkers over time | 51 months
  reporting the value of each biomarker at each patient's visit to visit
Describe and compare biomarkers according to clinical characteristics of participants | 51 months
  Value of each biomarker according to the clinical characteristics of participants
Describe changes in quality of life over time | 51 months
  Quality of life (SF-12 score) at each visit.
Describe changes in smoking habits over time | 51 months
  Smoking cessation rate achieved (partial and/or total) among participants active smokers
Describe changes in anxiety over time | 51 months
  anxiety (STAI-YA and STAI-YB) at each visit.
Describe and compare biomarkers according to medical characteristics of participants | 51 months
  Value of each biomarkers according to medical characteristics of participants
Describe and compare biomarkers according to geographic characteristics of participants | 51 months
  Value of each biomarkers according to geographic characteristics of participants
Describe and compare biomarkers according to socioeconomic characteristics of participants | 51 months
  Value of each biomarkers according to socioeconomic characteristics of participants

CONTACTS AND LOCATIONS:
Overall Officials: Mathilde LEFEVRE, Study Director — ASSISTANCEPUBLIQUE HOPTAUX DE MARSEILLE
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France